CLINICAL TRIAL: NCT01298206
Title: Case-control Study of Pandemic A/H1N1 Influenza Risk Factors In Lebanon
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: XPD10-150 PANFLU; CDRF-BEP-22033 (Other: Biosecurity Engagement Program, US Department of State)
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: A/H1N1 Influenza; Swine Flu
Keywords: A/H1N1 Influenza; swine flu; virus disease; Avian flu
MeSH Terms: conditions — Orthomyxoviridae Infections; Virus Diseases; Influenza in Birds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected from cases(ie positive for pandemic influenza by RT PCR) will be processed in order to isolate and characterize the viruses causing infection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- H1N1 not exposed controls: For every enrolled H1N1 case, the study will enroll 2 sex matched controls. On the date of enrollment of a case, 2 sex-matched controls will be located from the same clinic from which the case was enrolled. Enrolled controls will then be verified to be free from influenza infection at the time of enrollment by RT-PCR.
- H1N1 exposed Cases: A swab will be collected from cases to verify presence of pandemic influenza. Testing positive for influenza A/H1N1 by RT PCR to be enrolled will be confirmed as a case. The participant will be presented with a questionnaire that will capture exposure data through a group of variables assessing underlying health conditions, symptoms, use of influenza vaccine, travel, occupational setting, and other demographic variables. Cases will be contacted once during the study.

SUMMARY:
The pandemic A/H1N1 virus was named "swine flu" when the current outbreak started. Although it is not yet confirmed that the index case acquired the virus from pigs, the nomenclature "swine flu" was due to the fact that the virus is triple-reassortant with genes from swine, avian, and human influenza origins. A total of 57,809 cases were reported in the WHO EMRO region, 693 of whom have died (1.2% case fatality). Lebanon had 1,838 confirmed cases with 5 deaths, it is estimated that 4% of these cases required hospitalization. Most cases of pandemic influenza presented with fever, cough, and sore throat. Other common symptoms included myalgia, headache, and rhinorrhea. The pandemic A/H1N1 virus appears to be very successful at human-to-human transmission. It is also causing infections beyond the traditional seasonal variation of previous human influenza viruses. Unlike seasonal influenza viruses that usually cause severe infections requiring hospitalization among the elderly and children under 5 years old, the pandemic A/H1N1 viruses are causing more severe illness among young adults. Several reports have associated certain underlying conditions with severe illness. Such conditions were pregnancy, asthma, diabetes, obesity, and heart disease.

DETAILED DESCRIPTION:
This study will measure risk and protective factors associated with pandemic A/H1N1 infection. This study will also be able to estimate risk factors for severe illness requiring hospitalization or leading to death. These factors are: travel history, exposure to other confirmed or suspected cases, obesity, pregnancy, influenza vaccination history, residency in nursing homes, attendance of daycares, tobacco use, and other comorbidities (pulmonary diseases, cardiovascular diseases, diabetes, renal insufficiency). Unlike other descriptive studies, this analytical case-control study will enable to accurately measure the strength of association between potential risk factors and outcome. By isolating viruses from specimens collected from cases, this study will be able to characterize these viruses and document any genetic mutations or antiviral resistance.

The main objectives of this study are:

1. To investigate the risk factors of infection with the pandemic A/H1N1 viruses.
2. To characterize influenza viruses causing infection.
3. If enough severe cases were enrolled to make it statistically feasible, this study will investigate the risk factors of severe illness or death associated with infection with the pandemic A/H1N1 viruses.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to participate by signing a consent form/assent statement, and completing the study requirements.
* Be willing to provide nasal swab.
* Testing negative for influenza A/H1N1 by RT PCR to be enrolled as a control.
* Testing positive for influenza A/H1N1 by RT PCR to be enrolled as a case.

Exclusion Criteria:

* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy. (Note that this study has chosen to exclude such populations because of their increased risk of acquiring infections, they are relatively few, and are not representative of a national sample).

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases will be selected from the outpatient clinics and inpatient units at American Univeristy of Beirut thus the study team expect that selection bias would be minimal. Confirmed cases attending other healthcare facilities for whom contact information is available, will be contacted and invited to participate in this study. Controls will be selected from the outpatient clinics and inpatient units of the Internal Medicine, Family Medicine, and Pediatric and Adolescent Medicine Departments at AUBMC. Cases and controls attending the hospital will be from the same catchment area, thus coming from the same geographical areas, have similar socioeconomic status, and have similar chances of exposure to influenza viruses. Other influenza case control studies have matched on sex and enrolled hospital-based controls.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
This study will investigate the risk factors with pandemic A/H1N1 virus by measuring the degree of exposure to virus; | One (1) year
  This study hypothesize that certain factors make people more vulnerable to be infected with A/H1N1, such as traveling to H1N1 infected area, exposure to infected patients, no influenza vaccination, residency in nursing homes, attendance of daycares, poor health and etc.

SECONDARY OUTCOMES:
This study will characterize influenza viruses causing infection by using molecular and cultural techniques | One (1) year
  Through these techniques, the study will isolate and characterize influenza viruses causing infection and morbidity severity of infection among the enrolled cases.
This study will investigate the risk factors of severe illness or death associated with infection with the pandemic A/H1N1 viruses. | One (1) year
  This study hypothesizes that certain factors make patients infected with A/H1N1 more vulnerable to severe illness or death, such as obesity, pregnancy, tobacco use, and other co-morbidities (pulmonary diseases, cardiovascular diseases, diabetes, and renal insufficiency).

CONTACTS AND LOCATIONS:
Overall Officials: Ghazi Kayali, Ph.D, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- American University of Beirut, Beirut, Beyrouth, Lebanon

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org